CLINICAL TRIAL: NCT05162924
Title: Efficacy of Chiropractic Spinal Manipulative Therapy in Patients With Primary Chronic Low Back Pain: a Mechanistic Randomized Controlled Trial
Brief Title: Mechanisms of Chiropractic Spinal Manipulation for Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Real Centro Universitario Maria Cristina (Other)
Collaborators: Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz (Other); Université du Québec à Trois-Rivières (Other); University of Alcala (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SMTCLBP
Record Dates: First submitted 2021-12-02; First posted 2021-12-17 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Chronic Low-back Pain
Keywords: Chronic low back pain; Spinal manipulation; Central sensitization; Pressure pain thresholds; Cytokines; Chiropractic
MeSH Terms: interventions — Manipulation, Spinal

STUDY DESIGN:
Intervention Model Description: Randomized placebo-controlled trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Patients will be randomly allocated to either one of two groups receiving real or sham spinal manipulation. The outcomes assessors will be unaware of the group allocation. The investigator will be unaware of the outcomes measured in patients.
  Healthy participants in the control group will be unaware of any study hypothesis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Spinal manipulation (Experimental): Group receiving 12 sessions of spinal manipulative therapy in the lumbar area
  Interventions: Other: Spinal Manipulation
- Placebo (Placebo Comparator): Group receiving 12 sessions of placebo spinal manipulative therapy in the lumbar area
  Interventions: Other: Placebo
- Healthy controls (No Intervention): A healthy control population will receive no treatment during the same time period (4 weeks) to measure the same physiological variables and their evolution.

INTERVENTIONS:
Other: Spinal Manipulation — Manual therapy technique applied by a chiropractor in the form of a high-velocity low-amplitude force to the lumbopelvic spine
  Arms: Spinal manipulation
Other: Placebo — Placebo spinal manipulation consisting in the application by a chiropractor of a lower-velocity lower-amplitude force to gluteal muscles in a non-intentional direction
  Arms: Placebo

SUMMARY:
This is a mechanistic randomized controlled trial on the effects of chiropractic spinal manipulative therapy on patients with chronic low back pain. It is designed as a mechanistic trial, in which the main objective is to identify which variables related to central sensitization can help predict the response to spinal manipulation, and the evolution of which of these variables can help explain clinical changes in chronic low back pain patients receiving spinal manipulative therapy.

DETAILED DESCRIPTION:
The study is a mechanistic randomized controlled trials on the effects of chiropractic spinal manipulative therapy on patients with chronic low back pain. 100 chronic low back pain patients will be randomly allocated to receive 12 sessions over 4 weeks of spinal manipulative therapy or placebo spinal manipulation. The main objective is to identify variables related to a central sensitization or nociplastic pain phenotype can help predict the response to spinal manipulation. Additionally, changes in these variables during the treatment period will be used to identify potential pain mechanisms involved in pain relief by spinal manipulation. An additional group of 50 healthy volunteers will be used to measure the same variables and their evolution during 4 weeks in a healthy control population. Response to treatment will be measured according to changes in pain intensity and disability.

ELIGIBILITY:
Healthy volunteers will be accepted for that specific comparison group. Those volunteers must demonstrate no evidence of any systemic pathology, inflammatory, psychiatric, neurological or pain condition.

Inclusion Criteria:

* diagnosis of primary chronic low back pain (performed in the initial evaluation or previously received by a healthcare professional), with or without leg pain
* minimum of three months of duration

Exclusion Criteria:

* diagnosis of neuropathic pain in the lower extremity
* evidence of specific pathology affecting the lumbar spine
* diagnosis of psychiatric disorder or pain disorder affecting the hand/thumb or in the vicinity of the lumbar area
* intake corticosteroids, opioids or anticytokine medications
* pregnancy
* having been treated with spinal manipulation in the previous 12 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2021-12-17 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-01-15 (Actual)

PRIMARY OUTCOMES:
Pain intensity | 4 weeks
  Pain intensity will be measured by showing patients a numerical rating scale from 0 (no pain at all) to 100 (maximum possible pain), and patients will rate with a number their current pain, highest, lowest and average during the 7 previous days (baseline) or the days following the previous session.
Oswestry Low Back Pain Disability Index | 4 weeks
  The Oswestry Disability Index (ODI) questionnaire provides the level of self-reported disability in activities of daily living (ADL) related to low back pain. It includes 10 items rated on a Likert scale from 0-5. The total range of possible scores is from 0-50, where 0 means no disability at all, and 50 is the maximal disability.

SECONDARY OUTCOMES:
Pain Catastrophizing Scale | 4 weeks
  The Pain Catastrophizing Scale (PCS) provides the level of catastrophizing beliefs and emotions that a person has with regards to his/her own pain experience, in this case, low back pain. It includes 13 items rated on a Likert scale from 0-4. The total range of possible scores is from 0-52, where 0 is the lowest possible level of catastrophizing and 52 the highest. This scale will also be used in healthy participants.
Central Sensitization Inventory | 4 weeks
  The Central Sensitization Inventory (CSI) identifies key symptoms associated with central sensitization and provides a quantification for the degree of these symptoms, which help to identify a central sensitization phenotype patients with chronic pain. It includes 25 items rated on a Likert scale from 0-4. The total range of possible scores is from 0-100, where 0 is the lowest possible level of central sensitization symptoms and 100 the highest. Additionally, the CSI asks one more question related to the previous diagnosis of either one of 10 conditions that have been related to central sensitization. this part is informative and is not used for scoring purposes. This scale will also be used in healthy participants.
Pressure pain thresholds | 4 weeks
  Pressure pain thresholds (PPTs) are part of quantitative sensory testing. The aim is to identify the threshold and the sensitivity to suprathreshold pressure stimulation in different areas of the patients' bodies. A digital algometer will be used (Wagner Force Dial FPX, Greenwich, CT, USA) to measure PPTs in the lumbar segment of greatest pain for each patient (2cm lateral to the spinous process or the posterosuperior iliac spine if applicable) locally, in the dermatome of this segment in the lower limbs, at the regional level four segments cranial from the segment of greatest pain, and remotely at the level of the thenar eminences. Measures will always be taken bilaterally two times, and averaged. At that time, the patient will rate in a numerical rating scale from 0 to 100 the intensity of the first painful stimulation (suprathreshold sensitivity). For healthy participants, pressure pain thresholds will be measured at every segment of the lumbar spine and in the thenar eminences.
Urinary levels of cytokine Tumor Necrosis Factor alpha | 4 weeks
  Tumor Necrosis Factor alpha (TNF-a) is a pro-inflammatory cytokines that have been involved with different stages of low back pain. First morning urine samples will be taken from patients and healthy participants at the beginning and the end of the trial period. Samples will be stored at -20ºC and concentrations will be measured with a sandwich ELISA. TNF-a will be the only cytokine used for before and after changes.
Beck Depression Inventory II | 4 weeks
  The Beck Depression Inventory (BDI-II) identifies key symptoms associated with clinical depression and provides a quantification for the presence and severity of depressive symptoms. It includes 21 items rated on a Likert scale from 0-3. The total range of possible scores is from 0-63, where 0 is the lowest possible level of depressive symptoms and 63 the highest.This scale will also be used in healthy participants.
Generalized Anxiety Disorder scale | 4 weeks
  The Generalized Anxiety Disorder (GAD) identifies key symptoms associated with generalized anxiety disorder and provides a quantification for the presence and severity of these symptoms. It includes 7 items rated on a Likert scale from 0-3. The total range of possible scores is from 0-63, where 0 is the lowest possible level of depressive symptoms and 21 the highest. The threshold of 10/21 is used to diagnose generalized anxiety disorder. This scale will also be used in healthy participants.
Expectations of pain relief | 4 weeks
  Participants will rate in a numerical rating scale their expectations of pain relief at the end of the trial. It will consist on a scale from -100 (maximum reduction in current pain) to 0 (no change) to +100 (maximum imaginable pain increase).

OTHER OUTCOMES:
Pain frequency | Baseline measurement for exploratory purposes
  Chronic pain patients will describe whether their pain is episodic (pain-free periods of at least 4 week duration) or fluctuating (no pain-free periods of at least 4 week duration)
Pain duration | Baseline measurement for exploratory purposes
  Pain duration at baseline since the onset of low back pain, described in months
Pain widespreadness | Baseline measurement for exploratory purposes
  Patients will draw in a digital application (Symptom Mapper) the extent of their body affected by pain.
Pain in lower extremity | Baseline measurement and changes post-treatment for exploratory purposes
  The presence of pain in the lower extremity concomitant or related to low back pain will be recorded as Yes/No answer.
Pain medication use | Baseline measurement and changes post-treatment for exploratory purposes
  The use of pain medication (apart from the ones referred to in the exclusion criteria) will be reported as Yes/No answer, and a description will be noted.
Clinical criteria 1 for diagnosing central sensitization type of pain | Baseline measurement for exploratory purposes
  A set of clinical criteria (defined by Smart et al., Manual Therapy 2015 and Nijs et al., Pain Physician 2015) will be used to classify patients as having central sensitization pain, this first one will be answered with a "Yes" or "No" regarding whether their pain is disproportionate to damage to lumbar tissues.
Clinical criteria 2 for diagnosing central sensitization type of pain | Baseline measurement for exploratory purposes
  A set of clinical criteria will be used to classify patients as having central sensitization pain, this second one will be answered with a "Yes" or "No" regarding whether their pain has a diffuse anatomical distribution.
Sex | Baseline measurement for exploratory purposes
  Biological sex (Male or Female)
Age | Baseline measurement for exploratory purposes
  Age (measured in years)
Level of education | Baseline measurement for exploratory purposes
  Education level (3 categories: basic, high school or university level)
Chronic disease comorbidities | Baseline measurement for exploratory purposes
  The presence of other chronic disease comorbidities will be assessed as Yes/No answer.
Adverse reactions (type) | Will be collected at the beginning of every treatment session, except the first one
  Type of adverse reaction to treatment (muscle stiffness, increased pain, radiating discomfort, and others - described by the patient)
Adverse reactions (onset) | Will be collected at the beginning of every treatment session, except the first one
  Onset of adverse reaction to treatment (immediately, up to 24 hours, or more than 24 hours after the previous session)
Adverse reactions (duration) | Will be collected at the beginning of every treatment session, except the first one
  Duration of adverse reaction to treatment (minutes, hours (< 24 hours), 24-48 hours, or > 48 hours)
Adverse reactions (severity) | Will be collected at the beginning of every treatment session, except the first one
  Severity of adverse reaction to treatment (very mild, mild, moderate, severe, very severe)

CONTACTS AND LOCATIONS:
Overall Officials: Arantxa Ortega-De Mues, PhD, Principal Investigator — Real Centro Universitario María Cristina; Mathieu Piché, PhD, Principal Investigator — Université du Québec à Trois-Rivières
Locations (1):
- Real Centro Universitario María Cristina, El Escorial, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication will be shared
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD data will be available in 2022 or immediately after publication
Access Criteria: Data will be available upon request via email to the corresponding author of the publication

REFERENCES:
- [Background] Smart KM, Blake C, Staines A, Thacker M, Doody C. Mechanisms-based classifications of musculoskeletal pain: part 1 of 3: symptoms and signs of central sensitisation in patients with low back (+/- leg) pain. Man Ther. 2012 Aug;17(4):336-44. doi: 10.1016/j.math.2012.03.013. Epub 2012 Apr 23. PMID 22534654
- [Background] Nijs J, Apeldoorn A, Hallegraeff H, Clark J, Smeets R, Malfliet A, Girbes EL, De Kooning M, Ickmans K. Low back pain: guidelines for the clinical classification of predominant neuropathic, nociceptive, or central sensitization pain. Pain Physician. 2015 May-Jun;18(3):E333-46. PMID 26000680
- [Background] Shraim MA, Masse-Alarie H, Hodges PW. Methods to discriminate between mechanism-based categories of pain experienced in the musculoskeletal system: a systematic review. Pain. 2021 Apr 1;162(4):1007-1037. doi: 10.1097/j.pain.0000000000002113. PMID 33136983
- [Derived] Gevers-Montoro C, Ortega-De Mues A, Piche M. Mechanisms of chiropractic spinal manipulative therapy for patients with chronic primary low back pain: protocol for a mechanistic randomised placebo-controlled trial. BMJ Open. 2023 Feb 10;13(2):e065999. doi: 10.1136/bmjopen-2022-065999. PMID 36764718

DOCUMENTS (2):
  • Study Protocol (2021-12-15): https://cdn.clinicaltrials.gov/large-docs/24/NCT05162924/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-15): https://cdn.clinicaltrials.gov/large-docs/24/NCT05162924/SAP_001.pdf